CLINICAL TRIAL: NCT02281630
Title: Phase II, Randomized, Placebo-controlled, Double-blind, Parallel-group Study of KWA-0711 Administered Orally for 4 Weeks to Evaluate Its Efficacy and Safety, and to Determine Its Optimal Dose in Patients With Chronic Constipation (CC)
Brief Title: Phase II Dose-Finding Study of KWA-0711 in Patients With Chronic Constipation (CC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KWA1204
Record Dates: First submitted 2014-10-22; First posted 2014-11-03 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; CC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- KWA-0711 High dose (Experimental)
  Interventions: Drug: KWA-0711
- KWA-0711 Low dose (Experimental)
  Interventions: Drug: KWA-0711
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KWA-0711
  Arms: KWA-0711 High dose; KWA-0711 Low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KWA-0711, and to determine its optimal dose in Chronic Constipation (CC) patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who experienced fewer than three SBMs per week for more than 6 months prior to the enrollment.
* The patients who experienced one or more of the following signs or symptoms during more than 25% of bowel movements for more than 6 months: straining, lumpy or hard stools, and a sensation of incomplete evacuation.

Exclusion Criteria:

* Patients who have secondary constipation caused by systemic disorder.
* Patients who have organic constipation.
* Patients who received intestinal resection.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2015-04-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly number of Spontaneous Bowel Movements (SBMs) at Week 1 | 1 week

SECONDARY OUTCOMES:
Complete SBM (CSBM) frequency and responder rate | 4 weeks
SBM frequency and responder rate | 4 weeks
Time to first SBM after the initial dose | 4 weeks
Stool consistency | 4 weeks
Degree of straining | 4 weeks
Abdominal bloating and discomfort | 4 weeks
Use of rescue medications | 4 weeks
Global assessment of constipation severity | 4 weeks
Japanese version of IBS-QOL | 4 weeks
Global assessment of treatment effectiveness | 4 weeks
Satisfaction rating for the condition of bowel movements | 4 weeks
Adverse events, ECGs, vital signs, and clinical labs | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuro Takei, Study Director — Kissei Pharmaceutical Co., Ltd.
Locations (1):
- Tokyo and Other Japanese City, Japan

REFERENCES:
- [Derived] Fukudo S, Endo Y, Hongo M, Nakajima A, Abe T, Kobayashi H, Nakata T, Nakajima T, Sameshima K, Kaku K; Mizagliflozin Study Group. Safety and efficacy of the sodium-glucose cotransporter 1 inhibitor mizagliflozin for functional constipation: a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Gastroenterol Hepatol. 2018 Sep;3(9):603-613. doi: 10.1016/S2468-1253(18)30165-1. Epub 2018 Jul 25. PMID 30056028